CLINICAL TRIAL: NCT04008173
Title: The International Survey of Acute Coronary Syndromes-ARCHIVES
Acronym: ISACS-ARCHIVES
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Raffaele Bugiardini, Full Professor of Cardiology, University of Bologna
Other Study IDs: University of Bologna
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndrome; Unstable Angina Pectoris; Myocardial Infarction; Coronary Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Myocardial Infarction; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Databases with significant genomic data (e.g., genome-wide association studies, medical sequencing, molecular diagnostic assays), are expected to be deposited as well. Likewise, physical bio-samples can be included in the ISACS ARCHIVES.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Male: Non-interventional patient registry
  Interventions: Other: Non-interventional patient registry
- Female: Non-interventional patient registry
  Interventions: Other: Non-interventional patient registry
- Kidney Disease: Non-interventional patient registry
  Interventions: Other: Non-interventional patient registry
- Diabetes: Non-interventional patient registry
  Interventions: Other: Non-interventional patient registry
- Elderly: Non-interventional patient registry
  Interventions: Other: Non-interventional patient registry

INTERVENTIONS:
Other: Non-interventional patient registry — Non-interventional patient registry

SUMMARY:
ISACS ARCHIVES network is part of ISACS TC (NCT01218776) health care program. It is a collaborative network of research centers that support the rapid development of new scientific information and analytic tools. The ISACS ARCHIVES network assists health care providers, scientists, and policymakers seeking unbiased information about the outcomes, clinical effectiveness, safety, and appropriateness of health care items and services, particularly prescription medications and medical devices in acute coronary syndromes (ACS).

DETAILED DESCRIPTION:
Purpose

ISACS-TC investigators may deposit to the ISACS ARCHIVES their registry data acquired prior to the first submitted date of ISACS-TC at ClinicalTrials.gov (October 7, 2010). Non- ISACS investigators with ACS data are welcome to deposit their data to the ISACS ARCHIVES as well. In this case the data may have been acquired prior or later than October 7, 2010. The data in the ISACS ARCHIVES will be catalogued and made available to the general research community. The ISACS ARCHIVES will use an established informatics infrastructure, hosted and managed by the ISACS TC (NCT01218776) and the Department of Electrical and Computer Engineering, University of California, Los Angeles, California, which will enable the sharing and use of data. The NIH. Gov. Registration number for the ISACS ARCHIVES will serve as the key for ACS related data submissions to the contact persons.

Applicable Data The ISACS ARCHIVES will accept only de-identified data from human subjects' studies on ACS (for a definition of human subjects see: https://humansubjects.nih.gov/glossary). This will include data from clinical trials, epidemiological surveys, and other types of studies involving human subjects. Databases with significant genomic data (e.g., genome-wide association studies, medical sequencing, molecular diagnostic assays), are expected to be deposited as well. Likewise, physical bio-samples can be included in the ISACS ARCHIVES.

Data Sharing Procedures Data submitted to the ISACS ARCHIVES must be de-identified by the investigator prior to submission. Submitted data will be subjected to algorithms that check for basic data accuracy. Any problematic data items will be summarized in a report and returned to the investigator for corrective action, if necessary, before data are accepted. Data will be made available for sharing with general research community 2 months after the deposit. This 2-month embargo period will provide study investigators with protected time to check for basic data accuracy. After the embargo, the data will be made available for sharing with the general research community. Investigators will be able to gain access to ISACS ARCHIVES data by submitting a data access request to ISACS TC (NCT01218776) contact persons. Data requests will be reviewed by an ISACS ARCHIVES Data Access Committee. The Department of Electrical and Computer Engineering, University of California, Los Angeles, California will collect data.

ISACS Data Archive Sharing The following is a summary of tasks and expectations related to submitting data to the ISACS ARCHIVES. The purpose of this summary is to provide an overview of data submission and data sharing via the ISACS ARCHIVES. This list only provides a summary of tasks.

Investigators are expected to:

1. Collect Personally Identifiable Information (PII) from research subjects that will allow for the creation of the ISACS ARCHIVES Global Unique Identifier.
2. Provide a de-identified subject ID, which is required for submission of data to the ISACS ARCHIVES.
3. Complete and submit a Data-Sharing Agreement and Permission (DSAP) to ISACS TC (NCT01218776) contact persons.
4. Review the ISACS TC data definition for the measures/experiments expected and define the project's data definition harmonized to that standard.
5. Work with ISACS TC (NCT01218776) contact persons to define any undefined measures in accordance with ISACS TC practices.
6. Specify the expected measures to be collected by the project in a summary table to be forwarded to the ISACS TC (NCT01218776) contact persons.
7. Address any post submission quality assurance and quality control (QA/QC) checks that have been identified by the ISACS TC (NCT01218776).
8. Create an ISACS ARCHIVES Library, linking a result from a publication, pipeline, or discovery of the data sent to ISACS ARCHIVES to its records for publications of results.

Policy Implementation ISACS ARCHIVES expects investigators and their institutions to provide basic plans for policy implementation

At present PI Study Investigators:

* ISACS TC. International Survey of Acute Coronary Syndromes in Transitional Countries (ClinicalTrials.gov Identifier NCT01218776) from October 2010 to present. Contact person: Raffaele Bugiardini, MD University of Bologna email raffaele.bugiardini@unibo.it
* HORACS: hospital registry for acute coronary syndrome in Serbia from January 2002 to September 2010. Contact person: Zorana Vasiljevic, MD Medical Faculty, University of Belgrade, email zoranav@eunet.rs
* EMMACE-3 X. Long-term Follow-up of Health-Related Quality of Life in Patients With Acute Coronary Syndrome (ClinicalTrials.gov Identifier NCT01955525) during the period of 2011 to 2013. Contact person: Chris P Gale University of Leeds email c.p.gale@leeds.ac.uk

ISACS ARCHIVES Data Access Committee

* Raffaele Bugiardini, University of Bologna (Principal Investigator)
* Chris P Gale, University of Leeds
* Olivia Manfrini, University of Bologna
* Lina Badimon, Cardiovascular Research Institute (ICCC), CiberCV-Institute Carlos III, IIB-Sant Pau, Hospital de la Santa Creu i Sant Pau, Autonomous University of Barcelona
* Mihaela van der Schaar, University of Cambridge

ISACS ARCHIVES Data Sharing Coordinators

* Edina Cenko University of Bologna
* Jinsung Yoon, Department of Electrical and Computer Engineering, University of California, Los Angeles

Sponsor University of Bologna

Inquiries

Please direct all inquiries to:

Principal Investigator: Raffaele Bugiardini, MD University of Bologna

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndromes

Exclusion Criteria:

* under age or not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted with a diagnosis of acute coronary syndromes
Sampling Method: Probability Sample
Enrollment: 130000 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All causes death | 30 days
  All causes death
All causes death | 6 months
  All causes death
All causes death | 1 year
  All causes death

SECONDARY OUTCOMES:
Cardiovascular death | up to 1 year
  Cardiovascular death
Recurrent myocardial infarction | up to 1 year
  A disorder characterized by signs and symptoms related to acute ischemia of the myocardium secondary to coronary artery disease
Pharmacogenomics | up to 1 year
  DNA sequence data to predict drug response and to inform drug discovery and development
Cardiovascular genetics of coronary heart disease | up to 1 year
  Common variant genotyping for risk prediction

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Bugiardini, MD, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bugiardini R, Yoon J, Kedev S, Stankovic G, Vasiljevic Z, Milicic D, Manfrini O, van der Schaar M, Gale CP, Badimon L, Cenko E. Prior Beta-Blocker Therapy for Hypertension and Sex-Based Differences in Heart Failure Among Patients With Incident Coronary Heart Disease. Hypertension. 2020 Sep;76(3):819-826. doi: 10.1161/HYPERTENSIONAHA.120.15323. Epub 2020 Jul 13. PMID 32654558
- [Background] Bugiardini R, Cenko E, Yoon J, van der Schaar M, Kedev S, Gale CP, Vasiljevic Z, Bergami M, Milicic D, Zdravkovic M, Krljanac G, Badimon L, Manfrini O. Concerns about the use of digoxin in acute coronary syndromes. Eur Heart J Cardiovasc Pharmacother. 2022 Aug 11;8(5):474-482. doi: 10.1093/ehjcvp/pvab055. PMID 34251454
- [Background] Vasiljevic Z, Scarpone M, Bergami M, Yoon J, van der Schaar M, Krljanac G, Asanin M, Davidovic G, Simovic S, Manfrini O, Mickovski-Katalina N, Badimon L, Cenko E, Bugiardini R. Smoking and sex differences in first manifestation of cardiovascular disease. Atherosclerosis. 2021 Aug;330:43-51. doi: 10.1016/j.atherosclerosis.2021.06.909. Epub 2021 Jun 26. PMID 34233252
- [Derived] Bugiardini R, Yoon J, Mendieta G, Kedev S, Zdravkovic M, Vasiljevic Z, Milicic D, Manfrini O, van der Schaar M, Gale CP, Bergami M, Badimon L, Cenko E. Reduced Heart Failure and Mortality in Patients Receiving Statin Therapy Before Initial Acute Coronary Syndrome. J Am Coll Cardiol. 2022 May 24;79(20):2021-2033. doi: 10.1016/j.jacc.2022.03.354. PMID 35589164